CLINICAL TRIAL: NCT03078946
Title: Dexmedetomidine Versus Morphine and Midazolam in Prevention and Treatment of Delirium After Adult Cardiac Surgery; a Randomized, Double-blind Clinical Trial
Brief Title: Dexmedetomidine Versus Morphine and Midazolam in Prevention and Treatment of Delirium After Adult Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Lecturer of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1775
Record Dates: First submitted 2017-03-03; First posted 2017-03-14 (Actual); Results first posted 2020-08-28 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Delirium
Keywords: Cardiac surgery; delirium; dexmedetomidine; morphine; midazolam
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Morphine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (N=30) (Active Comparator)
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Morphine with Midazolam (N=30) (Active Comparator)
  Interventions: Drug: Morphine and Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — 30 patients received a loading dose of 1 μg/kg dexmedetomidine (Precedex; Hospira, Precedex 200 mcg/2 ml, Hospira. Inc, Lake Forest, USA) diluted in 100 ml 0.9% saline infused over 10 min immediately postoperative, followed by continuous infusion of 0.2- 0.7 μg/kg/h
  Arms: Dexmedetomidine Group (N=30)
Drug: Morphine and Midazolam — 30 patients received morphine in a dose of 10-50μg/ kg/hr as an analgesic (Morphine Sulphate ampoule; 10 mg/ 1ml, Misr Co.- Egypt) with midazolam in a dose of 0.05mg/kg up to 0.2 mg/kg (Dormicum; Roche; USA; ampoule containing 15 mg/3 ml mixed in sugar-free apple juice limiting the total volume mixed with a double volume of apple juice) repeated as needed.
  Arms: Morphine with Midazolam (N=30)

SUMMARY:
This randomized double-blind parallel clinical study was conducted on 60 patients undergoing elective cardiac surgery under general anesthesia, at least 60 yr old, ASA I and II, 70-100 kg body weight and height 160-180 cm. Patients were randomized to: group A=30 patients receiving dexmedetomidine infusion (0.4- 0.7 µg /kg/h) or group B= 30 patients receiving morphine in a dose of 10-50μg/kg/hr as an analgesic with midazolam in a dose of 0.05mg/kg up to 0.2 mg/kg repeated as needed. Titration of the study medications infusions was conducted to maintain light sedation (RASS) (-2 to +1). Primary outcome was the prevalence of delirium measured daily via Confusion Assessment Method for intensive care. If Delirium and agitation occurred: haloperidol 2.5-5 mg IV was given in repeated boluses. Secondary outcomes included ventilation time, additional sedation/analgesia, hemodynamics and adverse effects.

DETAILED DESCRIPTION:
Upon arrival at the ICU, a standardized protocol for postoperative care was implemented for all patients. Infusion rates for all sedative protocols were titrated in order to achieve and maintain light sedation (RASS -2 to +1) before extubation and (RASS 0) after extubation. All patients were extubated when deemed clinically appropriate according to local protocols. Because of their specific pharmacologic properties (i.e., respiratory depression), patients were weaned off propofol or midazolam infusions before extubation, whereas patients receiving dexmedetomidine were extubated while still on the medication and were kept on the maintenance infusion as deemed clinically necessary for a maximum of 24 hours.

Initial assessment and stabilization of both patient groups include; Clinical examination, hemodynamics (invasive blood pressure, heart rate, drains), activated clotting time, electrocardiography, chest x-ray and arterial blood gases including sodium and potassium. All patients were allowed to take 200 μg fentanyl and 5mg midazolam immediately on admission. Daily electrocardiography, chest x-ray, arterial blood gases including sodium and potassium, kidney function, coagulation profile if valve surgery or bleeding occurred, liver function if delirium occurred and CRP quantitative titre.

Delirium was monitored and reassessed up to a maximum of 7 days after surgery and the assessment takes place in two steps; Firstly, the level of consciousness must be assessed using the Richmond Agitation-Sedation Scale. If the patient appears to have a RASS score≥3, then evaluation of delirium using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) can be performed. The CAM-ICU includes the assessment of 4 different features; acute change or fluctuating course of mental status, inattention, altered level of consciousness and disorganized thinking. CAM-ICU is considered positive when features 1 and 2 and either 3 or 4 are present (11). The CAM-ICU was performed once daily before midday, independent of additional analgesia or sedation. Abnormal or delirious behavior was recorded every shift by the bedside nurse (nurse:patient ratio 1:1) and reviewed by the research team. The number of delirium days was determined by following delirious patients until 7 days after surgery. Patients were considered delirium-free when they were free of delirium for more than 24 h and alive.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery under general anesthesia
* at least 60 yr old
* ASA physical status I and II
* 70-100 kg body weight
* height 160-180 cm.

Exclusion Criteria:

* Patients with impaired kidney or liver functions
* history of cardiac or central nervous system disease
* uncontrolled medical disease (diabetes mellitus and hypertension)
* coagulation defect
* history of drug or alcohol abuse
* history of chronic pain or daily intake of analgesics
* history of intake of non-steroidal anti-inflammatory drugs or opioids within 24 h before surgery
* allergy to the used medications
* or patient's refusal

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

REFERENCES:
- [Result] Azeem TMA, Yosif NE, Alansary AM, Esmat IM, Mohamed AK. Dexmedetomidine vs morphine and midazolam in the prevention and treatment of delirium after adult cardiac surgery; a randomized, double-blinded clinical trial. Saudi J Anaesth. 2018 Apr-Jun;12(2):190-197. doi: 10.4103/sja.SJA_303_17. PMID 29628826
- See also: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5875204/ — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5875204/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were excluded if: (1) patient's refusal, (2) allergy to any drugs of the study, (3) history of drug or alcohol abuse, (4) history of uncontrolled diabetes or hypertension, (5) history of chronic pain or daily intake of analgesics within 24 h before surgery, and (6) impaired kidney or liver functions.
Period: Overall Study
Arm/Group | Dexmedetomidine Group (N=30) | Morphine With Midazolam (N=30)
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Group (N=30) | Morphine With Midazolam (N=30) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (4.8) | 66.7 (5.6) | 65.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 13 | 15 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Delirium (Number of Patients (in Digits))
Time Frame: Delirium was reported on day 7 post-surgery
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine Group (N=30) | Morphine With Midazolam (N=30)
Number analyzed (Participants) | 30 | 30
participants | 1 | 2

2. Primary Outcome: The C-reactive Protein (CRP) Quantitative Titer Daily as Part of the Routine Clinical Care as a Prognostic Factor for Delirium (mg/L)
Time Frame: The maximum serum CRP level during the ICU stay was designated as max-CRP on day 7 post-surgery
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dexmedetomidine Group (N=30) | Morphine With Midazolam (N=30)
Number analyzed (Participants) | 30 | 30
mg/L | 127.1 (253.29) | 101 (253.3)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine Group (N=30) | Morphine With Midazolam (N=30)
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/30
Other Adverse Events (participants affected / at risk) | 1/30 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine Group (N=30) (N=30) | Morphine With Midazolam (N=30) (N=30)
Delirium (Nervous system disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine Group (N=30) (N=30) | Morphine With Midazolam (N=30) (N=30)
Delirium (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No